CLINICAL TRIAL: NCT01416103
Title: Alcohol and Employment - a Randomized Controlled Trial
Brief Title: Alcohol and Employment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: TRYG Foundation (Other)
Responsible Party: Principal Investigator, Maja Bæksgaard Hansen, Research assistant, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 61110- 1986 (tryg, p7)
Record Dates: First submitted 2011-07-12; First posted 2011-08-12 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Alcohol Abuse
MeSH Terms: conditions — Alcoholism | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): Intervention group
  Interventions: Other: Intervention group
- Intervention control (Placebo Comparator): Control group
  Interventions: Other: Control group

INTERVENTIONS:
Other: Intervention group — Alcohol treatment paralleling welfare-to-work participation: The participants are referred to the municipalities' outpatient alcohol treatment programmes and at the same time referred to an ordinary welfare-to-work programme.
  Arms: Intervention group
Other: Control group — The participants will as usual be referred to the welfare-to-work schemes deemed most appropriate by the caseworker. The intervention is no different than what the municipality would have offered if the participant was not part of the study.
  Arms: Intervention control

SUMMARY:
The purpose of the study is to determine whether welfare-to-work schemes combined with alcohol treatment are more efficient than a welfare-to-work scheme alone, for unemployed citizens with alcohol problems.

DETAILED DESCRIPTION:
Background and purpose: The Tryg Foundation Denmark has awarded funds for a study that tests how to most efficiently combine welfare-to-work schemes with efforts against alcoholism, in relation to a return to the labour market.

The study will be carried out in a number of Danish municipalities in the time frame 2011-2014.

The purpose of the study is to determine whether a welfare-to-work scheme combined with alcohol treatment is more efficient than a welfare-to-work scheme alone, for unemployed citizens with alcohol problems.

Design: If the welfare recipient meets the inclusion criteria, then the recipient is provided with information about the project by the caseworker. If the recipient wishes to participate in the project he/she is asked to fill out a consent form and a questionnaire regarding employment status, alcohol consumption, other habits of abuse, health status and background information.

Welfare recipients who do not wish to participate will as usual be referred to the welfare-to-work schemes deemed most appropriate by the caseworker.

The intervention is designed as a randomized controlled trial, where heavy drinkers who meet the inclusion criteria and wish to participate will be allocated to either:

A) An intervention group receiving welfare-to-work scheme combined with alcohol treatment.

or

B) A control group receiving only welfare-to-work scheme.

After 6 and 12 months there will be a follow-up where participants will be asked to answer a questionnaire with questions about their employment status, alcohol consumption, other habits of abuse, health status and background information.

In this study ANCOVA is chosen to analyses the effective of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have an audit-score above 7.
* Participants must be unemployed and receive welfare-to-work schemes when included.

Exclusion Criteria:

* Participants who have an audit-score below 8.
* Participants who have a normal job.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2011-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the participant's employment status at 6 and 12 months. | 6 and 12 months
  Change in the participant's employment status, i.e. a) ordinary job, b) change in the participant transfer payments or in other ways approaching the labour market.
  Employment status is measured with self-reported questionnaires and with a number of administrative registers connected through each participant's personal identification number.

SECONDARY OUTCOMES:
Change from baseline in the participant's alcohol consumption, health status and readiness for the labour market at 6 and 12 months. | 6 and 12 months
  1. Alcohol consumption is measured with The Alcohol Use Disorder Test (AUDIT) and with the average volume of alcohol per week.
  2. Health status is measured with the standardized instrument EQ5D and with questionnaire on self rated health.
  3. Readiness for the labour market is measured with five self rated questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Morten Grønbæk, MD, PhD, Study Director — Centre for Intervention Research in Health Promotion and Disease Prevention
Locations (1):
- National Institute of Public Health - University of Southern Denmark, Copenhagen, Copenhagen K, Denmark

REFERENCES:
- [Derived] Hansen MB, Kloster S, Danquah IH, Nielsen AS, Becker U, Tjornhoj-Thomsen T, Tolstrup JS. "A welfare recipient may be drinking, but as long as he does as told--he may drink himself to death": a qualitative analysis of project implementation barriers among Danish job consultants. BMC Public Health. 2015 Mar 18;15:264. doi: 10.1186/s12889-015-1620-x. PMID 25886200